CLINICAL TRIAL: NCT04703153
Title: LIQUIK: LIQUId Biopsy for Detection of Actionable Genomic BiomarKers in Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Acronym: LIQUIK
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lucence Health Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LIQUIK-01
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: biomarkers; cell-free DNA; cfDNA; CGP; liquid biopsy; lung cancer; NGS; tissue biopsy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the non-inferiority of a cfDNA amplicon-based liquid biopsy technology vs. standard of care tissue biopsy-based NGS in detecting guideline- recommended biomarkers in patients with metastatic non-squamous Non-small Cell Lung Cancer (NSCLC), amongst other endpoints.

To explore the non-inferiority of cfDNA-based LiquidHALLMARK test vs. cfDNA-based liquid biopsy competitor, both qualitatively and quantitatively for actionable mutation (percentage of allele frequency) profile results in a population of subjects who have at least one actionable mutation detected by tissue biopsy.

DETAILED DESCRIPTION:
1. To explore the non-inferiority of a cfDNA amplicon-based liquid biopsy technology vs. standard of care tissue biopsy-based NGS in detecting guideline- recommended biomarkers in patients with metastatic non-squamous Non-small Cell Lung Cancer (NSCLC), amongst other endpoints.
2. To explore the non-inferiority of cfDNA-based LiquidHALLMARK test vs. cfDNA-based liquid biopsy competitor, both qualitatively and quantitatively for actionable mutation (percentage of allele frequency) profile results in a population of subjects who have at least one actionable mutation detected by tissue biopsy.
3. Condition or disease: NSCLC
4. Intervention/treatment: Observational

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed, histologically confirmed, metastatic non-squamous NSCLC whom:

   * Have already received standard-of-care tissue genotyping using Next Generation Sequencing (NGS) for lung cancer at clinician's discretion, including at least EGFR, ALK, RET, ROS1, NTRK fusions, MET, BRAF, HER2 and KRAS, in the last 90 (ninety) calendar days of enrollment or
   * Are scheduled to receive standard-of-care tissue genotyping using Next Generation Sequencing (NGS) for lung cancer at clinician's discretion, including at least EGFR, ALK, RET, ROS1, NTRK fusions, MET, BRAF, HER2 and KRAS.
2. Tissue genotyping is to be performed by Comprehensive Genomic Profiling (CGP) either in-house (at study site laboratory) or at an outside CAP-accredited laboratory by sending out tissue for analysis. Tissue CGP must be performed by Next Generation Sequencing (NGS). Other genomic platforms and methodologies for tissue genomic profiling, such as PCR, FISH or IHC are not eligible for this study.

   Eligible subjects whose physician intends to order tissue for genotyping at study enrollment, but there is insufficient material for analysis are still eligible for enrollment.
3. Patients with no previous surgical treatment, such as cancer resection, except patients with previously resected early stage NSCLC (stage I-IIIA), now with recurrent and metastatic disease, if tissue from a site of metastatic disease has been obtained within a 90 (ninety) calendar-day window of enrollment.
4. Treatment naïve patients for metastatic disease, i.e., no previous systemic therapy such as chemotherapy, targeted therapy or immunotherapy for metastatic disease. Adjuvant therapy is allowable for eligible patients who have received prior adjuvant molecularly targeted therapy and they have completed this therapy at least 6 weeks prior to study enrollment.
5. Patients with previously treated localized NSCLC (stage I-IIIA) are eligible if primary surgical resection and/or radiation treatment was completed at least 6 months prior to the development of metastatic disease and adjuvant chemotherapy, or targeted therapy completed at least 6 weeks prior to study enrollment.
6. No past history of any histologically confirmed malignant invasive neoplasm (excluding the current diagnosis of lung cancer and any non-melanoma skin cancer that was treated surgically with curative intent) in the last 3 years.
7. Ability to understand a written informed consent and willingness to sign it.
8. ≥ 21 years of age.

Exclusion Criteria:

1. Patients who are unwilling to follow-up for evaluation of response to therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naïve newly diagnosed, histologically confirmed, metastatic NSCLC patients
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the non-inferiority of cfDNA-based LiquidHALLMARK liquid biopsy assay vs. SOC tissue biopsy based NGS assay for mutation profile results | 34 months
  Explore the non-inferiority of cfDNA-based LiquidHALLMARK liquid biopsy assay vs. SOC tissue biopsy based NGS assay for mutation profile results in a population of subjects who have at least one of nine actionable genes (G9) - EGFR, ALK, RET, ROS1, NTRK fusions, MET, BRAF, ERBB2 and KRAS- detected by tissue biopsy.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - California Research Institute, Los Angeles, California
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Kaiser Permanente Hawaii Region Center for Integrated Health Care Research, Honolulu, Hawaii
  - University of Maryland - Marlene and Stewart Greenbaum Cancer Center, Baltimore, Maryland
  - New Jersey Cancer Care, Belleville, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Samol J, Ng D, Poh J, Tan MH, Dawar R, Carney J, Orsini J Jr, Scilla K, Tan YO, Chin TM, Toh CK, Goh BC, Lopes G. Prospective Multicenter Study Evaluating a Combined Circulating Tumor DNA and Circulating Tumor RNA Liquid Biopsy in Metastatic Non-Small Cell Lung Cancer (LIQUIK). JCO Precis Oncol. 2025 Jun;9:e2500181. doi: 10.1200/PO-25-00181. Epub 2025 Jun 26. PMID 40570258